CLINICAL TRIAL: NCT03677804
Title: Aortic Valve Reconstruction Using Autologous Pericardium: Single Center Experience With the OZAKI Technique
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00556; ch17Reuthebuch
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Aortic Valve Disease
Keywords: aortic valve reconstruction; OZAKI technique; autologous pericardium
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to analyse the short-term results of the first patients undergoing the OZAKI procedure (Aortic valve reconstruction using autologous pericardial tissue) at the department of cardiac surgery/ University Hospital Basel/ Switzerland.

DETAILED DESCRIPTION:
The reconstruction of the aortic valve using autologous pericardium, applying the technique Ozaki et al., published first in 2011 provides potential benefits due to the missing necessity of oral anticoagulation and its use in patients with small aortic annuli, because of the huge orifice area. There is a need of more data to evaluate the significance of this technique in the treatment of aortic valve stenosis and regurgitation. The department of cardiac surgery/ University Hospital Basel/ Switzerland started to use this technique in September 2015. The aim of this study is to analyse the short-term results of the first patients undergoing the OZAKI procedure.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve reconstruction using autologous Pericardium (OZAKI technique)

Exclusion Criteria:

* missing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing aortic valve reconstruction using autologous pericardium (OZAKI technique) in Universitätsspital Basel/ Switzerland since September 2015.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Change in aortic transvalvular gradient measured by transthoracic echocardiography | From Baseline (end of cardiac surgery) until 12 months after cardiac surgery
  Change in aortic transvalvular gradient ( to analyze aortic valve stenosis or insufficiency) measured by transthoracic echocardiography

SECONDARY OUTCOMES:
occurence of death | From Baseline (end of cardiac surgery) until 12 months after cardiac surgery
  Change in clinical Parameter: death
occurence of cardiac re-surgery | From Baseline (end of cardiac surgery) until 12 months after cardiac surgery
  Change in clinical parameter: cardiac re-surgery
occurence of stroke | From Baseline (end of cardiac surgery) until 12 months after cardiac surgery
  Change in clinical parameter: stroke

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Koechlin L, Schurr U, Miazza J, Imhof S, Maurer M, Erb J, Gahl B, Santer D, Berdajs D, Eckstein FS, Reuthebuch O. Echocardiographic and Clinical Follow-up After Aortic Valve Neocuspidization Using Autologous Pericardium. World J Surg. 2020 Sep;44(9):3175-3181. doi: 10.1007/s00268-020-05588-x. PMID 32458022